CLINICAL TRIAL: NCT03397589
Title: Coordinated Oral Health Promotion (CO-OP) Chicago
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Molly A. Martin, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-1090; UH3DE025483 (NIH)
Record Dates: First submitted 2017-12-22; First posted 2018-01-12 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Dental Caries in Children; Health Behavior; Healthcare Disparities
MeSH Terms: conditions — Health Behavior | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: cluster-randomized two arm trial with wait list control
Who Masked: Outcomes Assessor
Masking Description: Because of the nature of the intervention, participants will know after randomization which arm they are in. Outcomes assessors and data analysts will be masked to study arm. Most investigators will be masked to study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHW Arm (Experimental): The intervention is community health worker (CHW) services. CHWs trained in oral health will be assigned to half of the sites. Participants in these sites will be offered four in-person visits and follow-up phone calls over 12-months. These visits can occur at the location of the family's preference (recruitment site, home, or mutually-agreed upon other location). A core curriculum of oral health topics will be covered during visits, with an emphasis on developing and sustaining healthy oral health management routines for the entire family.
  Interventions: Behavioral: Community Health Worker (CHW) services
- Wait-list Control Arm (No Intervention): This arm will receive usual care. After completion of the final data collection at one year, participants and sites allotted to this arm will be offered CHW services.

INTERVENTIONS:
Behavioral: Community Health Worker (CHW) services — CHWs are non-clinical people who provide education, care coordination, and support to families.
  Arms: CHW Arm

SUMMARY:
This study assesses the impact of oral health promotion delivered by community health workers in medical clinics, Women, Infants and Children (WIC) centers, and family homes. Investigators will assess oral health behaviors in children aged 0 to 3.

DETAILED DESCRIPTION:
Dental caries is the most common chronic disease of childhood; an estimated 28% of children nationally aged 5 years and below have untreated dental disease. Pediatric dental caries are associated with pain, more severe infections, malnutrition, speech difficulties, poor school performance, cosmetic problems, and an overall lower quality of life. Similar to other chronic diseases, oral health disparities are seen with higher caries prevalence and worse outcomes in children from low income urban families and in children of African American and Latino ethnicity. These disparities have been demonstrated locally in Chicago. Many interventions have been implemented to attempt to reverse these disparities. Some involve public policy (fluorinated water), some are educational campaigns targeting individuals, while others focus on providing increased education and services through primary healthcare providers. Many of these programs have demonstrated efficacy but the disparities in oral health persist. The investigators propose this is because the interventions to date do not target the family as a whole and also have not targeted multiple levels simultaneously.

COordinated Oral health Promotion (CO-OP) Chicago brings together a team of clinical pediatricians and dentists, health researchers, and policy experts to rigorously test the ability of multiple oral health promotion interventions, both alone and in combination, to improve child and family oral health. The primary intervention is family-focused education and support from community health workers (CHWs). CO-OP Chicago will test the impact of a family-focused CHW intervention for oral health promotion when applied in clinical, community, and home settings. The primary study objective is to evaluate the efficacy of a one-year oral health CHW intervention, compared to usual care, to improve self-reported brushing frequency and observed plaque score in low income urban children under the age of 3 years old. The study's exploratory aim is to determine if the oral health CHW intervention impact on child tooth brushing behaviors varies when the CHWs are based out of a medical clinic compared to a community WIC center.

ELIGIBILITY:
Inclusion Criteria:

Caregiver:

* Provide a signed and dated informed consent form
* Age 18 or older
* Be the primary caregiver of a child age 6-36 months old. The primary caregiver is defined for this study as the person (or one of the people) who is consistently responsible for the child's daily routines and who is a legal guardian.
* If a child lives in multiple households, the caregiver must live with the child at least 5 days of the week.
* The child must be an active patient/client in the clinic/center where recruited.
* Speak English or Spanish
* Willing to comply with all study procedures and be available for the duration of the study

Child:

* Age 6-36 months old
* An active patient/client in the clinic/center where recruited
* A minimum of two fully erupted central maxillary incisors

Exclusion Criteria:

* Child with medical condition that limits his or her ability to conduct the study activities (such as severe developmental or cognitive delay, ventilator or oxygen dependence, oral aversion, severe facial deformities)
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study
* Anything that would place the research or intervention staff at increased risk

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - CEDA WIC Center Blue Island, Blue Island, Illinois
  - Chicago Department of Public Health WIC Centers (Greater Lawn Health Center, Friend Family Health Center, Westside Health Partnership), Chicago, Illinois
  - Mile Square Health Center (Main, Englewood, Cicero, South Shore, Back of the Yards), Chicago, Illinois
  - University of Illinois at Chicago Outpatient Care Center, Chicago, Illinois
  - Aunt Martha's Southeast Side Community Health Center, Chicago, Illinois
  - Vida Pediatrics, Chicago, Illinois
  - CEDA WIC Centers (Diversey, Irving Park), Chicago, Illinois
  - Aunt Martha's Pediatric Health & Wellness Center, Chicago Heights, Illinois
  - CEDA WIC Center Harvey, Harvey, Illinois
  - CEDA WIC Center Maywood, Maywood, Illinois
  - CEDA WIC Oak Park, Oak Park, Illinois
  - Aunt Martha's South Holland Community Health Center, South Holland, Illinois
  - CEDA WIC Summit, Summit, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Three years after the end of the CO-OP Chicago research activity, data will be publicly released. Data will be maintained by the study team, in partnership with the community clinical partner. Registration will be required to access or download data files. Registered users will receive technical assistance with questions or problems from the Methodology Research Core (MRC) at the University of Illinois at Chicago's Institute for Health Research and Policy or from the UCSF Coordinating Center. A data sharing agreement will be required that will describe the conditions and restrictions of their use; limited data access will be made available only to users who successfully complete a rigorous approval process by both the investigators and the community partners. Data sets will be encrypted for transfer to approved investigators.
Supporting Information: Study Protocol
Time Frame: These details are not fully developed.
Access Criteria: These details are not fully developed.

REFERENCES:
- [Derived] Martin MA, Avenetti D, Lee HH, Nordgren R, Berbaum ML, Edomwande Y, Cui L, Sandoval A. Community health worker intervention to improve tooth brushing in young children: Results from a cluster randomized controlled trial. Community Dent Oral Epidemiol. 2023 Jun;51(3):503-511. doi: 10.1111/cdoe.12768. Epub 2022 Jun 29. PMID 35766288
- [Derived] Martin MA, Zimmerman LJ, Rosales GF, Lee HH, Songthangtham N, Pugach O, Sandoval AS, Avenetti D, Alvarez G, Gansky SA. Design and sample characteristics of COordinated Oral health Promotion (CO-OP) Chicago: A cluster-randomized controlled trial. Contemp Clin Trials. 2020 May;92:105919. doi: 10.1016/j.cct.2019.105919. Epub 2019 Dec 30. PMID 31899372

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHW Arm | Wait-list Control Arm
Started | 211 | 209
Completed | 175 | 187
Not Completed | 36 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHW Arm | Wait-list Control Arm | Total
Number analyzed (Participants) | 211 | 209 | 420
Age, Continuous [Mean (Standard Deviation); unit: months] | 22.4 (6.8) | 20.8 (7.0) | 21.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 109 | 213
  Male | 107 | 100 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 115 | 111 | 226
  Not Hispanic or Latino | 96 | 98 | 194
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 92 | 84 | 176
  White | 21 | 36 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 98 | 89 | 187

OUTCOME MEASURES:

1. Primary Outcome: Parent-reported Tooth Brushing Frequency
Description: parents will be asked how often the child's teeth are brushed
Time Frame: 12-months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | CHW Arm | Wait-list Control Arm
Number analyzed (Participants) | 175 | 187
Participants
  Never brush | 1 | 1
  Sometimes, but not everyday brush | 12 | 15
  Once a day brush | 56 | 49
  Twice a day brush | 85 | 105
  More than twice a day brush | 21 | 17

2. Primary Outcome: Child Dental Plaque Score
Description: Disclosing solution is applied to child's teeth, images are taken, and plaque score is determined using the Oral health Index - Maxillary Incisor Score (OHI-MIS). The buccal surfaces of teeth #D, E, F, and G were scored from 0-3, with 3 being the worst (plaque on more than 2/3 of tooth surface) and 0 being the best (no plaque present). The four individual tooth scores (or less if child did not have four teeth) were then added and divided by the number of teeth for a final average score ranging from 0-3.
Time Frame: 12-months post-randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CHW Arm | Wait-list Control Arm
Number analyzed (Participants) | 161 | 160
score on a scale | 1.88 (0.64) | 1.85 (0.66)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each participant over a 1 year period, from enrollment through the 1 year data collection.
Arm/Group | CHW Arm | Wait-list Control Arm
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/209
Serious Adverse Events (participants affected / at risk) | 0/211 | 0/209
Other Adverse Events (participants affected / at risk) | 0/211 | 0/209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT03397589/Prot_SAP_ICF_000.pdf